CLINICAL TRIAL: NCT03002688
Title: OSUWMC EEI Sequential Cataract Patient Experience Project
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Deborah Lowery, Assistant Professor Clinical Anesthesiology, Ohio State University
Other Study IDs: 2016H0032
Record Dates: First submitted 2016-12-15; First posted 2016-12-26 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Cataract Surgery Experience
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sequential Cataract Surgery with Survey: Subjects eligible for the study will fall into the sequential cataract surgery group and be administered brief surveys.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Verbal survey will be given before and after the cataract surgery, and on the day following the second cataract surgery.

SUMMARY:
The purpose is to gauge the patients' level of comfort and anxiety for sequential cataract surgeries to assess if the second experience of cataract surgery differs from the initial experience.

DETAILED DESCRIPTION:
Each patient is scheduled to undergo two sequential cataract extractions under topical anesthesia with local anesthetic eye drops and minimal sedation- one on each eye. The surgeon, basic surgical procedure, anesthetic technique, and approximate length of procedure are reasonably similar and the patients act as their own control. Subjects in the study will answer very brief questions regarding anxiety and comfort about their surgery before and after each procedure, and on the day after their second surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing sequential cataract surgeries within a 6 week time period performed by the ophthalmologist, Amit Tandon, MD.
2. Aged 18 years and older.

Exclusion Criteria:

1. Cognitive impairment causing inability to participate in survey
2. Language barrier causing an inability to participate in survey
3. Healthcare POA or guardian leading to an inability to consent to survey
4. Physician autonomy; patients that are inappropriate for the study as deemed by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by their status presenting for surgery with one specific surgeon (A.T.) at the Eye and Ear Center at Gowdy Fields. Access will be through the preoperative anesthesia assessment performed by the attending anesthesiologist.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Pain | First and second cataract extraction surgery occuring within 6 weeks
  Pain will be evaluated using verbal survey after each cataract surgery, scheduled to occur within 6 weeks time; subject will be asked if there was any difference in pain between surgeries on the day after the second cataract surgery.
Anxiety | First and second cataract extraction surgery occuring within 6 weeks
  Anxiety will be evaluated using verbal survey before each cataract surgeries, scheduled to occur within 6 weeks time; subject will be asked if there was any difference in anxiety between surgeries on the day after the second cataract surgery.
Awareness | First and second cataract extraction surgery occuring within 6 weeks
  Awareness will be evaluated using verbal survey after each cataract surgeries, scheduled to occur within 6 weeks time; subject will be asked if there was any difference in awareness between surgeries on the day after the second cataract surgery.
Comfort Level | First and second cataract extraction surgery occuring within 6 weeks
  Comfort level will be evaluated using verbal survey after cataract surgeries, scheduled to occur within 6 weeks time; subject will be asked if there was any difference in comfort level between surgeries on the day after the second cataract surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Lowery, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No